CLINICAL TRIAL: NCT00281580
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, 4x4 Factorial Design Trial to Evaluate Telmisartan 20, 40 and 80 mg Tablets in Combination With Amlodipine 2.5, 5 and 10 mg Capsules After Eight Weeks of Treatment in Patients With Stage I or II Hypertension, With an ABPM Sub-study
Brief Title: Telmisartan (Micardis) and Amlodipine (Norvasc) - Factorial Design Study for the Treatment of Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1235.1; 2008-000874-19 (EudraCT Number: EudraCT)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2010-04-28 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Telmisartan

ARMS (16):
- Placebo (Placebo Comparator): Placebo once daily for eight weeks
  Interventions: Drug: Placebo
- Telmisartan 20 mg (Experimental): Telmisartan 20 mg once daily for eight weeks
  Interventions: Drug: Telmisartan 20 mg
- Telmisartan 40 mg (Experimental): Telmisartan 40 mg once daily for eight weeks
  Interventions: Drug: Telmisartan 40 mg
- Telmisartan 80 mg (Experimental): Telmisartan 80 mg once daily for eight weeks
  Interventions: Drug: Telmisartan 80 mg
- Amlodipine 2.5 mg (Experimental): Amlodipine 2.5 mg once daily for eight weeks
  Interventions: Drug: Amlodipine 2.5 mg
- Amlodipine 5 mg (Experimental): Amlodipine 5 mg once daily for eight weeks
  Interventions: Drug: Amlodipine 5 mg
- Amlodipine 10 mg (Active Comparator): Amlodipine 5 mg for two weeks and forced titrated to amlodipine 10 mg for six weeks once daily
  Interventions: Drug: Amlodipine 5 mg; Drug: Amlodipine 10 mg
- Telmisartan 20 / Amlodipine 2.5 (Experimental): Telmisartan 20/ Amlodipine 2.5 mg once daily for eight weeks
  Interventions: Drug: Telmisartan 20 mg; Drug: Amlodipine 2.5 mg
- Telmisartan 20 / Amlodipine 5 (Experimental): Telmisartan 20 / Amlodipine 5 mg once daily for eight weeks
  Interventions: Drug: Telmisartan 20 mg; Drug: Amlodipine 5 mg
- Telmisartan 20 / Amlodipine 10 (Experimental): Telmisartan 20 / Amlodipine 5 for two weeks and forced titrated to amlodipine 10 mg for six weeks
  Interventions: Drug: Amlodipine 10 mg; Drug: Telmisartan 20 mg; Drug: Amlodipine 5 mg
- Telmisartan 40 / Amlodipine 2.5 (Experimental): Telmisartan 40 / Amlodipine 2.5 for eight weeks
  Interventions: Drug: Amlodipine 2.5 mg; Drug: Telmisartan 40 mg
- Telmisartan 40 / Amlodipine 5 (Experimental): Telmisartan 40 / Amlodipine 5 for eight weeks
  Interventions: Drug: Amlodipine 5 mg; Drug: Telmisartan 40 mg
- Telmisartan 40 / Amlodipine 10 (Experimental): Telmisartan 40 / Amlodipine 5 for two weeks and forced titrated to amlodipine 10 mg for six weeks
  Interventions: Drug: Telmisartan 40 mg; Drug: Amlodipine 10 mg; Drug: Amlodipine 5 mg
- Telmisartan 80 / Amlodipine 2.5 (Experimental): Telmisartan 80 / Amlodipine 2.5 for eight weeks
  Interventions: Drug: Amlodipine 2.5 mg; Drug: Telmisartan 80 mg
- Telmisartan 80 / Amlodipine 5 (Experimental): Telmisartan 80 / Amlodipine 5 mg for eight weeks
  Interventions: Drug: Telmisartan 80 mg; Drug: Amlodipine 5 mg
- Telmisartan 80 / Amlodipine 10 (Experimental): Telmisartan 40 / Amlodipine 5 for two weeks and forced titrated to amlodipine 10 mg for six weeks
  Interventions: Drug: Amlodipine 5 mg; Drug: Telmisartan 80 mg; Drug: Amlodipine 10 mg

INTERVENTIONS:
Drug: Amlodipine 5 mg — Amlodipine 5 mg once daily for two weeks
  Arms: Telmisartan 80 / Amlodipine 10
Drug: Placebo — Placebo to Telmisartan and Amlodipine once daily for eight weeks
  Arms: Placebo
Drug: Telmisartan 20 mg — Telmisartan 20 mg once daily for eight weeks
  Arms: Telmisartan 20 mg
Drug: Telmisartan 40 mg — Telmisartan 40 mg once daily for eight weeks
  Arms: Telmisartan 40 / Amlodipine 10
Drug: Amlodipine 10 mg — Amlodipine 10 mg once daily for six weeks
  Arms: Telmisartan 20 / Amlodipine 10
Drug: Telmisartan 20 mg — Telmisartan 20 mg once daily for eight weeks
  Arms: Telmisartan 20 / Amlodipine 2.5
Drug: Telmisartan 80 mg — Telmisartan 80 mg once daily for eight weeks
  Arms: Telmisartan 80 / Amlodipine 10
Drug: Amlodipine 10 mg — Amlodipine 10 mg once daily for six weeks
  Arms: Telmisartan 80 / Amlodipine 10
Drug: Telmisartan 20 mg — Telmisartan 20 mg once daily for eight weeks
  Arms: Telmisartan 20 / Amlodipine 10
Drug: Amlodipine 5 mg — Amlodipine 5 mg once daily for two weeks
  Arms: Telmisartan 20 / Amlodipine 10
Drug: Amlodipine 5 mg — amlodipine 5g once daily for eight weeks
  Arms: Amlodipine 5 mg
Drug: Telmisartan 20 mg — Telmisartan 20 mg once daily for eight weeks
  Arms: Telmisartan 20 / Amlodipine 5
Drug: Amlodipine 5 mg — Amlodipine 5 mg once daily for eight weeks
  Arms: Telmisartan 40 / Amlodipine 5
Drug: Amlodipine 5 mg — amlodipine 5mg once daily for eight weeks
  Arms: Telmisartan 20 / Amlodipine 5
Drug: Amlodipine 2.5 mg — Amlodipine 2.5 mg once daily for eight weeks
  Arms: Amlodipine 2.5 mg
Drug: Amlodipine 2.5 mg — Amlodipine 2.5 mg once daily for eight weeks
  Arms: Telmisartan 80 / Amlodipine 2.5
Drug: Amlodipine 10 mg — Amlodipine 10 mg once daily for six weeks
  Arms: Telmisartan 40 / Amlodipine 10
Drug: Amlodipine 2.5 mg — Amlodipine 2.5 mg once daily for eight weeks
  Arms: Telmisartan 40 / Amlodipine 2.5
Drug: Telmisartan 80 mg — Telmisartan 80 mg once daily for eight weeks
  Arms: Telmisartan 80 mg
Drug: Telmisartan 80 mg — Telmisartan 80 mg once daily for eight weeks
  Arms: Telmisartan 80 / Amlodipine 5
Drug: Amlodipine 5 mg — Amlodipine 5 mg once daily for two weeks
  Arms: Telmisartan 40 / Amlodipine 10
Drug: Amlodipine 2.5 mg — Amlodipine 2.5 mg once daily for eight weeks
  Arms: Telmisartan 20 / Amlodipine 2.5
Drug: Telmisartan 40 mg — Telmisartan 40 mg once daily for eight weeks
  Arms: Telmisartan 40 / Amlodipine 2.5
Drug: Telmisartan 40 mg — Telmisartan 40 mg once daily for eight weeks
  Arms: Telmisartan 40 / Amlodipine 5
Drug: Amlodipine 5 mg — amlodipine 5g once daily for two weeks
  Arms: Amlodipine 10 mg
Drug: Amlodipine 5 mg — Amlodipine 5 mg once daily for eight weeks
  Arms: Telmisartan 80 / Amlodipine 5
Drug: Telmisartan 40 mg — Telmisartan 40 mg once daily for eight weeks
  Arms: Telmisartan 40 mg
Drug: Telmisartan 80 mg — Telmisartan 80 mg once daily for eight weeks
  Arms: Telmisartan 80 / Amlodipine 2.5
Drug: Amlodipine 10 mg — Amlodipine 10 mg once daily for six weeks
  Arms: Amlodipine 10 mg

SUMMARY:
To demonstrate that Micardis and Norvasc when used together are more effective at lowering blood pre ssure.

ELIGIBILITY:
Inclusion criteria:

Main Inclusion Criteria: Male and female patients >=18 years of age with Stage I or II hypertension defined as: a mean seated cuff diastolic blood pressure >=95 and <=119 mmHg Main

Exclusion criteria:

Exclusion Criteria:

1. Patient is pregnant; breast-feeding; unwilling to use birth control during the study; has secondary hypertension; severe renal dysfunction; hepatic insufficiency; stroke within the last six months; myocardial infarction, cardiac surgery, percutaneous transluminal coronary angioplasty, unstable angina or coronary artery bypass graft within the past three months; unstable or uncontrolled diabetes for the past three months defined as a glucosylates hemoglobin (HbA1c) greater than ten percent ; history of angioedema or hypersensitivity related to either study drug.
2. Systolic Blood Pressure (SBP) is greater than or equal to 180 millimeters of mercury (mmHg), Diastolic Blood Pressure (DBP) is greater than or equal to 110 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1461 (Actual)
Dates: Start 2006-04; Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (136):
- United States (101):
  - 1235.1.457 Boehringer Ingelheim Investigational Site, Fairhope, Alabama
  - 1235.1.368 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1235.1.389 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1235.1.411 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1235.1.429 Boehringer Ingelheim Investigational Site, Chandler, Arizona
  - 1235.1.420 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 1235.1.391 Boehringer Ingelheim Investigational Site, Cudahy, California
  - 1235.1.444 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 1235.1.445 Boehringer Ingelheim Investigational Site, Encino, California
  - 1235.1.357 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1235.1.465 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1235.1.441 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1235.1.409 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1235.1.406 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1235.1.414 Boehringer Ingelheim Investigational Site, Santa Ana, California
  - 1235.1.383 Boehringer Ingelheim Investigational Site, Spring Valley, California
  - 1235.1.395 Boehringer Ingelheim Investigational Site, Tustin, California
  - 1235.1.453 Boehringer Ingelheim Investigational Site, Milford, Connecticut
  - 1235.1.394 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 1235.1.354 Boehringer Ingelheim Investigational Site, Cooper City, Florida
  - 1235.1.451 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1235.1.372 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1235.1.396 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1235.1.390 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1235.1.430 Boehringer Ingelheim Investigational Site, Kissimmee, Florida
  - 1235.1.351 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 1235.1.398 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 1235.1.405 Boehringer Ingelheim Investigational Site, Mirimar, Florida
  - 1235.1.352 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1235.1.369 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1235.1.397 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1235.1.449 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1235.1.355 Boehringer Ingelheim Investigational Site, Rockledge, Florida
  - 1235.1.407 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1235.1.380 Boehringer Ingelheim Investigational Site, Tucker, Georgia
  - 1235.1.438 Boehringer Ingelheim Investigational Site, Gurnee, Illinois
  - 1235.1.373 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1235.1.375 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1235.1.415 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1235.1.412 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 1235.1.435 Boehringer Ingelheim Investigational Site, Arkansas City, Kansas
  - 1235.1.379 Boehringer Ingelheim Investigational Site, Lenexa, Kansas
  - 1235.1.421 Boehringer Ingelheim Investigational Site, Newtown, Kansas
  - 1235.1.356 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1235.1.423 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1235.1.387 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1235.1.424 Boehringer Ingelheim Investigational Site, Bay City, Michigan
  - 1235.1.385 Boehringer Ingelheim Investigational Site, Florissant, Missouri
  - 1235.1.452 Boehringer Ingelheim Investigational Site, Florissant, Missouri
  - 1235.1.365 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1235.1.431 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1235.1.454 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1235.1.426 Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - 1235.1.434 Boehringer Ingelheim Investigational Site, Stratford, New Jersey
  - 1235.1.366 Boehringer Ingelheim Investigational Site, East Syracuse, New York
  - 1235.1.377 Boehringer Ingelheim Investigational Site, Northport, New York
  - 1235.1.427 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1235.1.381 Boehringer Ingelheim Investigational Site, Williamsville, New York
  - 1235.1.410 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1235.1.400 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1235.1.422 Boehringer Ingelheim Investigational Site, Greenboro, North Carolina
  - 1235.1.403 Boehringer Ingelheim Investigational Site, Lenior, North Carolina
  - 1235.1.376 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1235.1.392 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1235.1.384 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1235.1.458 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1235.1.374 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1235.1.446 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1235.1.413 Boehringer Ingelheim Investigational Site, Marion, Ohio
  - 1235.1.359 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1235.1.361 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1235.1.436 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1235.1.448 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1235.1.386 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1235.1.439 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1235.1.440 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1235.1.408 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 1235.1.404 Boehringer Ingelheim Investigational Site, Lansdale, Pennsylvania
  - 1235.1.428 Boehringer Ingelheim Investigational Site, Penndel, Pennsylvania
  - 1235.1.370 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1235.1.433 Boehringer Ingelheim Investigational Site, Beaufort, South Carolina
  - 1235.1.462 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1235.1.417 Boehringer Ingelheim Investigational Site, Cordova, Tennessee
  - 1235.1.459 Boehringer Ingelheim Investigational Site, Jackson, Tennessee
  - 1235.1.363 Boehringer Ingelheim Investigational Site, New Tazewell, Tennessee
  - 1235.1.382 Boehringer Ingelheim Investigational Site, Selmer, Tennessee
  - 1235.1.442 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1235.1.399 Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - 1235.1.460 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1235.1.443 Boehringer Ingelheim Investigational Site, Georgetown, Texas
  - 1235.1.416 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1235.1.402 Boehringer Ingelheim Investigational Site, Lake Jackson, Texas
  - 1235.1.432 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 1235.1.456 Boehringer Ingelheim Investigational Site, Odessa, Texas
  - 1235.1.418 Boehringer Ingelheim Investigational Site, Plano, Texas
  - 1235.1.455 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 1235.1.358 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1235.1.464 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1235.1.437 Boehringer Ingelheim Investigational Site, Burke, Virginia
  - 1235.1.447 Boehringer Ingelheim Investigational Site, Fredericksburg, Virginia
  - 1235.1.371 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Argentina (6):
  - 1235.1.001 Boehringer Ingelheim Investigational Site, BsAs
  - 1235.1.004 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1235.1.005 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1235.1.006 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1235.1.002 Boehringer Ingelheim Investigational Site, Carlos Paz
  - 1235.1.003 Boehringer Ingelheim Investigational Site, Córdoba
- Brazil (5):
  - 1235.1.115 Universidade Federal do Pará, Belém
  - 1235.1.102 Liga de Hipertensão Arterial, Goiânia
  - 1235.1.101 Clínica Médica, Rio de Janeiro
  - 1235.1.103 Unidade de Hipertensão - ICHC -, São Paulo
  - 1235.1.109 Centro de Pesquisas do Hospital do Rim e Hipertensão, São Paulo
- Mexico (10):
  - 1235.1.203, Col. Magdalena de Las Salinas
  - 1235.1.210 Consultorio Privado, Durango, Durango
  - 1235.1.202, Guadalajara, Jalisco
  - 1235.1.209 Boehringer Ingelheim Investigational Site, Guadalajara, Jalisco
  - 1235.1.204, Lomas de Guevara, Guadalajara
  - 1235.1.208 "Ignacio Chávez", Mexico City
  - 1235.1.211 Obesidad Y Prevencion de Enfermedades, Mexico City
  - 1235.1.212 en Factores de riesgo cardiovascular, México
  - 1235.1.205 Fraccionamiento Industrias, San Luis Potosí City
  - 1235.1.207, Zapopan, Jalisco
- South Africa (14):
  - 1235.1.314 Boehringer Ingelheim Investigational Site, Benoni
  - 1235.1.302 Boehringer Ingelheim Investigational Site, Boksburg
  - 1235.1.306 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.1.309 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.1.310 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.1.311 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.1.304 Boehringer Ingelheim Investigational Site, Durban
  - 1235.1.312 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1235.1.313 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1235.1.307 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1235.1.303 Boehringer Ingelheim Investigational Site, Lenasia
  - 1235.1.305 Boehringer Ingelheim Investigational Site, Lenasia
  - 1235.1.301 Boehringer Ingelheim Investigational Site, Pretoria
  - 1235.1.308 Boehringer Ingelheim Investigational Site, Pretoria

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Pl): placebo tablet plus encapsulated placebo tablet, QD in morning
- Telmisartan 20 mg (T20): Telmisartan 20mg tablet, QD in morning
- Telmisartan 40 mg (T40): Telmisartan 40mg tablet, QD in morning
- Telmisartan 80 mg (T80): Telmisartan 80mg tablet, QD in morning
- Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5): T20mg tab plus encapsulated A2.5mg capsule, QD in morning
- Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5): T20mg tab plus encapsulated A5mg capsule, QD in morning
- Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10): T20mg tab plus 2 encapsulated A5mg capsule, QD in morning
- Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5): T40mg tab plus encapsulated A2.5mg capsule, QD in morning
- Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5): T40mg tab plus encapsulated A5mg capsule, QD in morning
- Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10): T40mg tabl plus 2 encapsulated A5mg capsule, QD in morning
- Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5): T80mg tab plus encapsulated A2.5mg capsule, QD in morning
- Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5): T80mg tab plus encapsulated A5mg capsule, QD in morning
- Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10): T80mg tab plus 2 encapsulated A5mg capsule, QD in morning
- Amlodipine 2.5 mg (A2.5): encapsulated Amlodipine 2.5 mg capsule, QD in morning
- Amlodipine 5 mg (A5): encapsulated Amlodipine 5 mg capsule, QD in morning
- Amlodipine 10 mg (A10): 2 encapsulated Amlodipine 5 mg capsule, QD in morning
Period: Overall Study
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Started | 46 | 42 | 130 | 135 | 44 | 46 | 44 | 47 | 143 | 129 | 48 | 146 | 142 | 50 | 140 | 129
Completed | 39 | 41 | 125 | 118 | 40 | 43 | 39 | 46 | 135 | 117 | 44 | 136 | 129 | 43 | 133 | 116
Not Completed | 7 | 1 | 5 | 17 | 4 | 3 | 5 | 1 | 8 | 12 | 4 | 10 | 13 | 7 | 7 | 13
Not completed — Adverse Event | 2 | 0 | 2 | 4 | 1 | 0 | 1 | 0 | 1 | 6 | 0 | 5 | 8 | 2 | 3 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 4 | 1 | 1 | 2 | 2 | 1 | 5
Not completed — Lack of Efficacy | 2 | 1 | 1 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Randomised in error; pregnancy; moving | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Treated set including all 1461 patients who were randomised to receive double-blind treatment and took at least one dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10) | Total
Number analyzed (Participants) | 46 | 42 | 130 | 135 | 44 | 46 | 44 | 47 | 143 | 129 | 48 | 146 | 142 | 50 | 140 | 129 | 1461
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (12.3) | 53.6 (10.4) | 52 (11) | 53.1 (11.3) | 54 (10.8) | 54.4 (10.2) | 51 (11.2) | 50.7 (10.2) | 52.3 (11.9) | 53.3 (11.3) | 54.8 (9.7) | 52.7 (11.9) | 53.9 (11.6) | 55.3 (10.4) | 53.1 (10.6) | 53.4 (10.7) | 53.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 64 | 75 | 18 | 25 | 18 | 21 | 72 | 67 | 26 | 72 | 78 | 23 | 68 | 64 | 724
  Male | 29 | 26 | 66 | 60 | 26 | 21 | 26 | 26 | 71 | 62 | 22 | 74 | 64 | 27 | 72 | 65 | 737

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean Diastolic Blood Pressure (DBP) (Observed Telmisartan Effect)
Description: Observed results
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (Last Observation Carried Forward (LOCF))
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic diastolic blood pressure measurement following treatment with target therapy (FAS-TC).
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Telmisartan 0 mg (T0): Overall: including Pl, A2.5, A5, and A10 treated groups
- Telmisartan 20 mg (T20): Overall: including all treatment groups involving T20
- Telmisartan 40 mg (T40): Overall: including all treatment groups involving T40
- Telmisartan 80 mg (T80): Overall: including all treatment groups involving T80
Arm/Group | Telmisartan 0 mg (T0) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80)
Number analyzed (Participants) | 355 | 171 | 440 | 457
mmHg | -13 (8.8) | -16.4 (7.8) | -16.2 (8.9) | -16.9 (8.6)

2. Primary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean DBP (Adjusted Telmisartan Effects)
Description: Results stem from an ANCOVA including the main effects of treatment with telmisartan, treatment with amlodipine, and country/region with baseline DBP included as a covariate.
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 0 mg (T0) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80)
Number analyzed (Participants) | 355 | 171 | 440 | 457
mmHg | -12.5 (0.5) | -16.8 (0.6) | -16.6 (0.4) | -17.2 (0.4)

3. Primary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean DBP (Observed Amlodipine Effects)
Description: Observed results
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Amlodipine 10 mg (A10): monotherapy (A5 titrated to A10)
Arm/Group | Placebo (Pl) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 349 | 185 | 466 | 423
mmHg | -12.3 (9.7) | -14.9 (8.8) | -15.6 (8.1) | -18.6 (7.7)

4. Primary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean DBP (Adjusted Amlodipine Effects)
Description: as for outcome 2
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 349 | 185 | 466 | 423
mmHg | -12.2 (0.5) | -15.3 (0.6) | -16.2 (0.4) | -19.3 (0.4)

5. Primary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean DBP (Observed Treatment Effects)
Description: Observed results
Time Frame: End-of-study visit (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 46 | 42 | 129 | 132 | 44 | 45 | 40 | 47 | 141 | 123 | 46 | 143 | 136 | 48 | 137 | 124
mmHg | -5.9 (9.4) | -13.2 (9) | -13.1 (10.1) | -13.6 (8.7) | -18 (7.8) | -15.7 (6.5) | -18.7 (7) | -16.2 (8.2) | -16 (7.6) | -19.6 (7.9) | -15.3 (7.5) | -17.8 (8.5) | -19.6 (7.9) | -10.4 (9.9) | -13 (7.9) | -16.5 (7.1)

6. Primary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean DBP (Adjusted Treatment Effects)
Description: as for outcome 2
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 46 | 42 | 129 | 132 | 44 | 45 | 40 | 47 | 141 | 123 | 46 | 143 | 136 | 48 | 137 | 124
mmHg | -6.2 (1.2) | -13.8 (1.3) | -13.4 (0.7) | -14 (0.7) | -18.3 (1.2) | -15.9 (1.2) | -19.3 (1.3) | -16.9 (1.2) | -16.5 (0.7) | -20.2 (0.7) | -15.7 (1.2) | -18.2 (0.7) | -20.1 (0.7) | -10.6 (1.2) | -13.4 (0.7) | -17.11 (0.7)

7. Primary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean DBP (Adjusted Treatment Effects, Excluding Pl)
Description: as for outcome 2
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic diastolic blood pressure measurement following treatment with target therapy (FAS-TC), excluding patients treated with placebo
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 42 | 129 | 132 | 44 | 45 | 40 | 47 | 141 | 123 | 46 | 143 | 136 | 48 | 137 | 124
mmHg | -13.8 (1.2) | -13.4 (0.7) | -14 (0.7) | -18.3 (1.2) | -15.9 (1.2) | -19.3 (1.3) | -16.9 (1.2) | -16.5 (0.7) | -20.2 (0.7) | -15.7 (1.2) | -18.2 (0.7) | -20.1 (0.7) | -10.6 (1.2) | -13.4 (0.7) | -17.1 (0.7)

8. Secondary Outcome: Change From Baseline at 8 Weeks in Seated Trough Cuff Mean Systolic Blood Pressure (SBP)
Description: Results stem from an ANCOVA including the main effects of treatment with telmisartan, treatment with amlodipine, and country/region with baseline SBP included as a covariate.
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic Systolic Blood Pressure measurement following treatment with target therapy (FAS-TC)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 46 | 42 | 129 | 132 | 44 | 45 | 40 | 47 | 141 | 123 | 46 | 143 | 136 | 48 | 137 | 124
mmHg | -2.5 (1.8) | -15.1 (1.9) | -14.6 (1.1) | -14.3 (1.1) | -18.8 (1.9) | -21 (1.9) | -24.4 (2) | -21.9 (1.8) | -21.8 (1.1) | -24.7 (1.1) | -17.4 (1.8) | -22.1 (1) | -26.4 (1.1) | -11.4 (1.8) | -15.4 (1.1) | -20.7 (1.1)

9. Secondary Outcome: Change From Baseline at 8 Weeks in Standing Trough Cuff Mean DBP
Description: as for outcome 2
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 46 | 42 | 128 | 129 | 44 | 45 | 40 | 47 | 139 | 123 | 46 | 142 | 134 | 46 | 137 | 122
mmHg | -4.9 (1.2) | -10.4 (1.3) | -10 (0.8) | -11.1 (0.8) | -14.9 (1.3) | -13.1 (1.3) | -16.9 (1.3) | -15.8 (1.2) | -13.6 (0.7) | -18.4 (0.8) | -13.4 (1.2) | -16.2 (0.7) | -19 (0.7) | -8.1 (1.2) | -11.3 (0.7) | -14.6 (0.8)

10. Secondary Outcome: Change From Baseline at 8 Weeks in Standing Trough Cuff Mean SBP
Description: as for outcome 8
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 46 | 42 | 128 | 129 | 44 | 45 | 40 | 47 | 139 | 123 | 46 | 142 | 134 | 46 | 137 | 122
mmHg | -0.5 (1.9) | -13.2 (2) | -13.2 (1.1) | -12.9 (1.1) | -17.4 (1.9) | -18.9 (1.9) | -22.3 (2) | -20.3 (1.8) | -20 (1.1) | -22.8 (1.1) | -17.4 (1.9) | -21.2 (1.1) | -24.9 (1.1) | -9.1 (1.9) | -14.7 (1.1) | -19.1 (1.2)

11. Other Pre Specified Outcome: Change From Baseline at 2,4,6,and 8 Weeks in Seated Trough Cuff DBP
Description: Observed results for key combination therapies
Time Frame: Baseline to nominal week over the trial
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 137 | 121 | 139 | 135
mmHg
  Week 2 | -14.5 (8.76) | -14.4 (7.62) | -15.3 (7.87) | -14.6 (6.76)
  Week 4 (N=133, 115, 135, 129) | -16.0 (7.24) | -18.1 (8.52) | -17.2 (7.56) | -18.8 (7.06)
  Week 6 (N=134, 118, 131, 124) | -17.1 (8.59) | -19.0 (8.30) | -18.0 (8.02) | -20.0 (8.18)
  Week 8 (N=133, 112, 132, 121) | -16.3 (7.42) | -19.5 (8.03) | -18.3 (8.28) | -20.0 (7.61)

12. Secondary Outcome: DBP Control
Description: DBP control is defined as DBP < 90 mmHg - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 141 | 123 | 143 | 136
percentage of participants | 71.6 | 82.1 | 74.8 | 85.3

13. Secondary Outcome: DBP Response
Description: DBP response is defined as DBP < 90 mmHg or a reduction of DBP of >= 10 mmHg - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 141 | 123 | 143 | 136
percentage of participants | 80.9 | 91.9 | 88.8 | 91.2

14. Secondary Outcome: SBP Response
Description: SBP Response is defined as SBP < 140 mmHg or a reduction of SBP of >= 10 mmHg - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 139 | 123 | 142 | 134
percentage of participants | 91.5 | 96.7 | 87.4 | 94.9

15. Other Pre Specified Outcome: BP Control
Description: Percentage of responders (SBP<140 mmHg and DBP<90 mmHg) for all patients - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic diastolic and systolic blood pressure measurement following treatment with target therapy (FAS-TC).
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 141 | 123 | 143 | 136
percentage of participants | 58.9 | 75.6 | 65.7 | 76.5

16. Secondary Outcome: BP Normality
Description: No: Mean seated SBP >=140 and/or mean seated DBP >=90 mmHg at trough High normal: mean seated SBP >=130 and <140 mmHg and mean seated DBP >=85 and <90 mmHg at trough Normal: mean seated SBP >=120 and <130 mmHg and mean seated DBP >=80 and <85 mmHg at trough Optimal: mean seated SBP < 120 mmHg and mean seated DBP <80 mmHg at trough
  - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic Systolic and Diastolic Blood Pressure measurement following treatment with target therapy (FAS-TC)
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 139 | 123 | 142 | 134
percentage of participants
  No (SBP>=140 and/or DBP>=90) | 41.1 | 24.4 | 34.3 | 23.5
  High Normal (140>SBP>=130 and 90>DBP>=85) | 28.4 | 30.1 | 30.1 | 22.1
  Normal (130>SBP>=120 and 85>DBP>=80) | 21.3 | 32.5 | 25.9 | 39.7
  Optimal (SBP<120 and DBP<80) | 9.2 | 13 | 9.8 | 14.7

17. Secondary Outcome: Change From Baseline in ABPM Hourly Mean (Relative to Dosing) DBP
Description: Observed results - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: FAS-ABPM: all patients of the FAS that participated in the ambulatory blood pressure monitoring (ABPM) sub-study and had a successful APBM at both baseline and following treatment with target therapy.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 57 | 57 | 56 | 52
mmHg
  Hour 1 | -10.7 (9.5) | -15.4 (11.6) | -12.7 (9.9) | -13.4 (9.7)
  Hour 2 | -9.8 (11.7) | -15 (12.2) | -13.4 (9.5) | -14.6 (12.4)
  Hour 3 | -11.2 (13.2) | -14.1 (12.6) | -14.8 (11.6) | -15.4 (12)
  Hour 4 | -11.3 (11.8) | -16.5 (13.2) | -15.6 (11.7) | -15.8 (10.8)
  Hour 5 | -13.1 (11) | -14.1 (14.4) | -16.3 (14.3) | -15.7 (10.9)
  Hour 6 | -10.9 (11.6) | -14.5 (12.4) | -14.6 (9.9) | -16.4 (11)
  Hour 7 | -12.8 (10.2) | -15.6 (13.9) | -12.9 (10.4) | -15.7 (14)
  Hour 8 | -12.1 (12.3) | -17.4 (13.6) | -12.7 (13.6) | -17.1 (12.9)
  Hour 9 | -13.1 (10.3) | -15.7 (14.4) | -14.3 (14.3) | -17.2 (13.8)
  Hour 10 | -11.8 (10.3) | -13.8 (13.5) | -14.7 (15.7) | -18.5 (12.9)
  Hour 11 | -11.2 (12.9) | -14.4 (11.9) | -15.1 (13.1) | -16.1 (12.8)
  Hour 12 | -12 (11.3) | -13.3 (12.9) | -12.5 (14.8) | -15.7 (12.2)
  Hour 13 | -10.3 (11.7) | -14.7 (14.3) | -14.1 (13.5) | -15.1 (10.6)
  Hour 14 | -8.9 (13.2) | -14.8 (14.1) | -13.4 (13.4) | -11 (14.9)
  Hour 15 | -10.3 (16) | -11.5 (14.3) | -11.9 (14.8) | -10 (12.7)
  Hour 16 | -10.1 (15) | -10.3 (15.4) | -11.3 (12) | -12.2 (13.6)
  Hour 17 | -9.8 (13.7) | -10.4 (14.4) | -11.2 (12.5) | -11.5 (13.1)
  Hour 18 | -11.9 (15) | -9.9 (12.4) | -10.3 (12.3) | -12.2 (11.9)
  Hour 19 | -9.1 (10.9) | -10.5 (13.7) | -11.9 (10.4) | -13.2 (11.3)
  Hour 20 | -11 (11.9) | -9.9 (12.4) | -12.6 (11.1) | -15.9 (11.1)
  Hour 21 | -10.4 (13) | -8.9 (13.2) | -8.5 (12.7) | -14.8 (9.7)
  Hour 22 | -11.1 (12.6) | -9.8 (13.7) | -9.7 (12.9) | -15.4 (9.9)
  Hour 23 | -9.8 (11.3) | -13.3 (13.4) | -9.9 (12.2) | -14.6 (9.4)
  Hour 24 | -11.1 (9.5) | -12.6 (11.5) | -12 (13.1) | -13.1 (11.9)

18. Secondary Outcome: Change From Baseline in ABPM Hourly Mean (Relative to Dosing) SBP
Description: Observed results - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 57 | 57 | 56 | 52
mmHg
  Hour 1 | -18.7 (12.9) | -20.2 (16.5) | -19.1 (13.4) | -17.5 (15.9)
  Hour 2 | -13.1 (16.5) | -22.0 (17.9) | -20.5 (16.6) | -21.9 (15.9)
  Hour 3 | -15.3 (16.1) | -17.9 (18.9) | -21.1 (17.8) | -22.4 (16.8)
  Hour 4 | -18.0 (16.9) | -24.4 (20.6) | -22.5 (16.5) | -23.8 (15.9)
  Hour 5 | -19.3 (13.6) | -21.1 (19.8) | -25.3 (18.1) | -24.0 (16.5)
  Hour 6 | -14.1 (14.0) | -22.6 (14.9) | -21.6 (15.9) | -24.6 (14.8)
  Hour 7 | -17.8 (14.5) | -24.3 (19.5) | -19.9 (17.7) | -22.4 (15.6)
  Hour 8 | -18.8 (17.1) | -24.1 (20.8) | -20.3 (18.6) | -21.8 (15.5)
  Hour 9 | -20.3 (15.6) | -24.9 (20.0) | -22.0 (19.2) | -25.6 (16.1)
  Hour 10 | -20.0 (16.0) | -22.9 (19.2) | -22.5 (19.3) | -26.8 (19.3)
  Hour 11 | -18.7 (17.4) | -20.9 (19.8) | -23.2 (16.7) | -24.9 (15.7)
  Hour 12 | -18.4 (16.8) | -20.3 (19.5) | -19.7 (19.1) | -25.0 (17.3)
  Hour 13 | -18.5 (16.9) | -21.7 (23.5) | -22.7 (18.3) | -24.7 (14.6)
  Hour 14 | -16.7 (17.6) | -21.6 (20.8) | -21.7 (19.2) | -20.2 (16.9)
  Hour 15 | -15.7 (18.1) | -19.4 (20.5) | -19.0 (20.2) | -18.9 (15.1)
  Hour 16 | -17.0 (16.9) | -17.7 (20.0) | -18.0 (16.0) | -19.8 (15.4)
  Hour 17 | -17.3 (17.3) | -17.9 (20.3) | -14.7 (15.8) | -19.1 (15.5)
  Hour 18 | -17.5 (18.6) | -17.4 (16.4) | -15.1 (16.8) | -19.6 (16.6)
  Hour 19 | -16.5 (15.6) | -19.7 (18.4) | -16.9 (15.3) | -20.9 (17.3)
  Hour 20 | -17.8 (16.4) | -18.0 (17.4) | -16.5 (15.3) | -24.4 (14.3)
  Hour 21 | -17.5 (15.9) | -17.8 (17.6) | -15.7 (16.4) | -22.7 (15.0)
  Hour 22 | -16.2 (15.9) | -15.7 (17.0) | -15.5 (18.7) | -23.8 (13.8)
  Hour 23 | -14.4 (14.6) | -18.9 (16.1) | -16.5 (19.1) | -22.4 (14.0)
  Hour 24 | -15.8 (14.9) | -20.7 (16.3) | -18.5 (18.1) | -19.9 (13.9)

19. Secondary Outcome: Change From Baseline in ABPM 24-hour Mean DBP
Description: Observed results - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 57 | 57 | 56 | 52
mmHg | -11 (7.2) | -13.2 (7.7) | -12.8 (7.4) | -14.6 (6.9)

20. Secondary Outcome: Change From Baseline in ABPM 24-hour Mean SBP
Description: Observed results - key combination therapies
Time Frame: End-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 57 | 57 | 56 | 52
mmHg | -17.3 (10.4) | -20.5 (13.9) | -19.5 (11.6) | -22.4 (9.8)

21. Secondary Outcome: Orthostatic Change in Trough Cuff Mean DBP
Description: Calculated as seated minus standing for all patients - key combination therapies
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 133 | 112 | 132 | 121
mmHg | 2.2 (5.7) | 1.7 (5.4) | 2 (5.4) | 1.1 (4.9)

22. Secondary Outcome: Orthostatic Change in Trough Cuff Mean SBP
Description: Calculated as seated minus standing for all patients - key combination therapies
Time Frame: Week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 133 | 112 | 132 | 121
mmHg | 0 (7.5) | 0.6 (8) | 0.9 (7.5) | 0.8 (7.3)

23. Primary Outcome: Change From Baseline in Seated Trough Cuff Mean DBP (Observed Telmisartan Effect)
Description: Observed results
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic diastolic blood pressure measurement following treatment with target therapy and were identified as having moderate or severe hypertension at baseline (FAS-TC-MS).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 0 mg (T0) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80)
Number analyzed (Participants) | 256 | 129 | 334 | 331
mmHg | -13.1 (9) | -16.8 (8) | -16.9 (8.9) | -17.7 (8.8)

24. Primary Outcome: Change From Baseline in Seated Trough Cuff Mean DBP (Adjusted Telmisartan Effects)
Description: as for outcome 2
Time Frame: Baseline to end-of-study (up to 8 weeks) visit (LOCF)
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 256 | 129 | 334 | 331
mmHg | -12.7 (0.5) | -17.3 (0.7) | -17.3 (0.5) | -18 (0.5)

25. Primary Outcome: Change From Baseline in Seated Trough Cuff Mean DBP (Observed Amlodipine Effects)
Description: Observed results
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Amlodipine 0 mg (A0) - Overall: Overall: including Pl, T20, T40, and T80 treatment groups
- Amlodipine 2.5 mg (A2.5) - Overall: Overall: including all treatment groups involving A2.5
- Amlodipine 5 mg (A5) - Overall: Overall: including all treatment groups involving A5
- Amlodipine 10 mg (A10) - Overall: Overall: including all treatment groups involving A10
Arm/Group | Amlodipine 0 mg (A0) - Overall | Amlodipine 2.5 mg (A2.5) - Overall | Amlodipine 5 mg (A5) - Overall | Amlodipine 10 mg (A10) - Overall
Number analyzed (Participants) | 257 | 137 | 349 | 307
mmHg | -12.7 (10.1) | -16 (8.4) | -16.3 (8.3) | -19.2 (7.8)

26. Primary Outcome: Change From Baseline in Seated Trough Cuff Mean DBP (Adjusted Amlodipine Effects)
Description: as for outcome 2
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Amlodipine 0 mg (A0) - Overall | Amlodipine 2.5 mg (A2.5) - Overall | Amlodipine 5 mg (A5) - Overall | Amlodipine 10 mg (A10) - Overall
Number analyzed (Participants) | 257 | 137 | 349 | 307
mmHg | -12.5 (0.5) | -16.4 (0.7) | -16.7 (0.5) | -19.7 (0.5)

27. Primary Outcome: Change From Baseline in Seated Trough Cuff Mean DBP (Observed Treatment Effects)
Description: Observed results
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 35 | 33 | 100 | 89 | 34 | 34 | 28 | 30 | 108 | 96 | 36 | 106 | 100 | 37 | 101 | 83
mmHg | -5.5 (10.1) | -13.9 (9.4) | -13.8 (10.2) | -13.9 (9.2) | -18.4 (7.9) | -15.8 (6.4) | -19.5 (7.2) | -18.7 (7.9) | -16.8 (7.5) | -19.6 (8.3) | -16.3 (7.7) | -18.8 (9) | -20.4 (7.3) | -11.4 (8.3) | -13.1 (8.1) | -17.1 (7.6)

28. Primary Outcome: Change From Baseline in Seated Trough Cuff Mean DBP (Adjusted Treatment Effects)
Description: as for outcome 2
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 35 | 33 | 100 | 89 | 34 | 34 | 28 | 30 | 108 | 96 | 36 | 106 | 100 | 37 | 101 | 83
mmHg | -5.8 (1.4) | -14.4 (1.4) | -14.2 (0.8) | -14.1 (0.9) | -18.9 (1.4) | -15.9 (1.4) | -19.7 (1.6) | -18.8 (1.5) | -17.2 (0.8) | -20.1 (0.8) | -16.6 (1.4) | -19.1 (0.8) | -21 (0.8) | -11.7 (1.4) | -13.3 (0.8) | -17.6 (0.9)

29. Primary Outcome: Change From Baseline in Seated Trough Cuff Mean DBP (Adjusted Treatment Effects, Excluding Pl)
Description: as for outcome 2
Time Frame: Up to 8 weeks (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic diastolic blood pressure measurement following treatment with target therapy and were identified as moderate or severe hypertension at baseline (FAS-TC-MS), excluding patients treated with placebo
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 33 | 100 | 89 | 34 | 34 | 28 | 30 | 108 | 96 | 36 | 106 | 100 | 37 | 101 | 83
mmHg | -14.5 (1.4) | -14.2 (0.8) | -14.1 (0.9) | -18.9 (1.4) | -15.9 (1.4) | -19.7 (1.5) | -18.8 (1.5) | -17.2 (0.8) | -20.1 (0.8) | -16.6 (1.4) | -19.1 (0.8) | -21 (0.8) | -11.7 (1.3) | -13.3 (0.8) | -17.6 (0.9)

30. Secondary Outcome: Change From Baseline in Seated Trough Pulse Rate
Description: Observed results for all patients - key combination therapies
Time Frame: End-of-study visit (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff Pulse Rate measurements included all treated patients that had at least one Pulse Rate measurement following treatment with target therapy (FAS-TC)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 141 | 123 | 143 | 136
bpm | 0 (8.8) | 0 (9.5) | 2.4 (9.3) | -1.5 (9.7)

31. Secondary Outcome: Change From Baseline in Seated Trough Cuff Mean SBP
Description: as for outcome 8
Time Frame: Up to 8 weeks (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic Systolic Blood Pressure measurement following treatment with target therapy and were identified as having moderate or severe hypertension at baseline (FAS-TC-MS)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 35 | 33 | 100 | 89 | 34 | 34 | 28 | 30 | 108 | 96 | 36 | 106 | 100 | 37 | 101 | 83
mmHg | -1.9 (2.1) | -15.6 (2.1) | -15.4 (1.2) | -15.4 (1.3) | -19 (2.1) | -22.1 (2.1) | -25.2 (2.3) | -23.2 (2.2) | -22.2 (1.2) | -25.3 (1.3) | -17.4 (2) | -22.5 (1.2) | -26.5 (1.2) | -12.4 (2) | -14.8 (1.2) | -21 (1.4)

32. Secondary Outcome: Change From Baseline in Standing Trough Cuff Mean DBP
Description: as for outcome 2
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10): T40mg tab plus 2 encapsulated A5mg capsule, QD in morning
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 35 | 33 | 99 | 86 | 34 | 34 | 28 | 30 | 107 | 96 | 36 | 105 | 100 | 35 | 101 | 81
mmHg | -4.2 (1.4) | -11.7 (1.5) | -10.9 (0.9) | -11.3 (0.9) | -15.1 (1.4) | -13.3 (1.4) | -17.6 (1.6) | -17.5 (1.5) | -14.2 (0.8) | -18 (0.9) | -14.5 (1.4) | -17.3 (0.8) | -19.2 (0.8) | -8 (1.4) | -11 (0.8) | -15.5 (0.9)

33. Other Pre Specified Outcome: Change From Baseline in Seated Trough Cuff DBP
Description: Observed results for mod-sev patients - key combination therapies
Time Frame: Nominal week over the trial
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 105 | 94 | 104 | 100
mmHg
  Week 2 | -14.7 (8.9) | -14.7 (7.8) | -16.1 (7.9) | -14.9 (6.7)
  Week 4 (N=102, 90, 102, 96) | -16.5 (6.8) | -18.2 (9.2) | -17.8 (7.6) | -19.2 (6.8)
  Week 6 (N=102, 92, 98, 96) | -17.9 (7.8) | -19.7 (8.7) | -18.9 (8.2) | -19.5 (8.4)
  Week 8 (N=102, 87, 99, 88) | -17.1 (7.4) | -19.4 (8.5) | -19.3 (8.7) | -21.1 (7.1)

34. Secondary Outcome: Change From Baseline in Standing Trough Cuff Mean SBP
Description: as for outcome 8
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 31
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Pl) | Telmisartan 20 mg (T20) | Telmisartan 40 mg (T40) | Telmisartan 80 mg (T80) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Number analyzed (Participants) | 35 | 33 | 99 | 86 | 34 | 34 | 28 | 30 | 107 | 96 | 36 | 105 | 100 | 35 | 101 | 81
mmHg | 1 (2.1) | -13.7 (2.1) | -13.6 (1.2) | -14 (1.3) | -16.2 (2.1) | -19.4 (2.1) | -23.2 (2.3) | -21.8 (2.2) | -20.4 (1.2) | -22.8 (1.3) | -16.3 (2) | -21.9 (1.2) | -24.3 (1.2) | -10.1 (2.1) | -13.2 (1.2) | -19.3 (1.4)

35. Secondary Outcome: DBP Control
Description: DBP control is defined as DBP < 90 mmHg - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 108 | 96 | 106 | 100
percentage of participants | 69.4 | 77.1 | 68.9 | 85

36. Secondary Outcome: DBP Response
Description: DBP response is defined as DBP < 90 mmHg or a reduction of DBP of >= 10 mmHg - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 108 | 96 | 106 | 100
percentage of participants | 81.5 | 89.6 | 87.7 | 93

37. Other Pre Specified Outcome: BP Control
Description: Responders SBP<10 mmHg and DBP<90 mmHg) for mod-sev patients - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic diastolic and systolic blood pressure measurement following treatment with target therapy and were identified as having moderate or severe hypertension at baseline (FAS-TC-MS).
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 108 | 96 | 106 | 100
percentage of participants | 53.7 | 70.8 | 58.5 | 77

38. Secondary Outcome: SBP Response
Description: SBP Response is defined as SBP < 140 mmHg or a reduction of SBP of >= 10 mmHg - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 108 | 96 | 106 | 100
percentage of participants | 88.9 | 96.9 | 84.9 | 95

39. Secondary Outcome: BP Normality
Description: as for outcome 16
Time Frame: Up to 8 weeks (LOCF)
Population: The full analysis set relating to the in-clinic trough cuff blood pressure measurements included all treated patients that had at least one in-clinic Systolic and Diastolic Blood Pressure measurement following treatment with target therapy and were identified as having moderate or severe hypertension at baseline (FAS-TC-MS)
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 108 | 96 | 106 | 100
percentage of participants
  No (SBP>=140 and/or DBP>=90) | 46.3 | 29.2 | 41.5 | 23
  High Normal (140>SBP>=130 and 90>DBP>=85) | 25.9 | 29.2 | 26.4 | 27
  Normal (130>SBP>=120 and 85>DBP>=80) | 18.5 | 30.2 | 21.7 | 41
  Optimal (SBP<120 and DBP<80) | 9.3 | 11.5 | 10.4 | 9

40. Secondary Outcome: Change From Baseline in ABPM Hourly Mean (Relative to Dosing) DBP
Description: Observed results for mod-sev patients - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 108 | 96 | 106 | 100
mmHg
  Hour 1 | -11 (10.8) | -16.9 (10.8) | -13.8 (10.1) | -13.7 (10.3)
  Hour 2 | -8.8 (12.3) | -16.3 (12.5) | -13.9 (9.3) | -15.9 (13)
  Hour 3 | -11.2 (14.4) | -13.8 (11.2) | -16.4 (11.3) | -16.1 (11.7)
  Hour 4 | -10.7 (12.4) | -16.3 (13.6) | -15.9 (11.8) | -16.8 (11.3)
  Hour 5 | -12.8 (10.5) | -15.3 (14.3) | -17.2 (14.3) | -16.6 (10.9)
  Hour 6 | -10.5 (12.2) | -15.3 (12.6) | -15.2 (10.1) | -16.3 (11.8)
  Hour 7 | -13.8 (11.1) | -15.3 (11.4) | -12.9 (10.9) | -17.5 (14.6)
  Hour 8 | -13.3 (13.1) | -19.4 (13.7) | -13.5 (14.2) | -17.8 (13.7)
  Hour 9 | -14 (11) | -16.6 (14.2) | -15.8 (14.3) | -18.1 (14.1)
  Hour 10 | -10.7 (11.1) | -14.6 (14) | -17 (14.2) | -20.8 (13.2)
  Hour 11 | -11.4 (13.9) | -14.8 (12.6) | -16.8 (10.5) | -17.9 (12.9)
  Hour 12 | -12.4 (12.2) | -13.9 (12.4) | -14.3 (12.2) | -16.6 (12.9)
  Hour 13 | -9.7 (13) | -14.9 (14.5) | -14.1 (12.5) | -15.9 (10.9)
  Hour 14 | -8.5 (14.3) | -14.5 (14.6) | -15.1 (11.2) | -12 (14.6)
  Hour 15 | -10.5 (16.6) | -10.5 (13.6) | -13.8 (14.7) | -10 (12.9)
  Hour 16 | -10.9 (15) | -10.3 (16.3) | -12.8 (12.2) | -13.7 (13)
  Hour 17 | -10.1 (14.1) | -9.8 (14.9) | -11.5 (12.5) | -12.3 (10.8)
  Hour 18 | -11.8 (15.6) | -9.9 (13.5) | -10.6 (10.3) | -12.8 (10.8)
  Hour 19 | -9 (11.7) | -11.6 (13.9) | -12.2 (10.6) | -12.5 (11.8)
  Hour 20 | -10 (12.3) | -10.9 (13.1) | -13.3 (11.2) | -15.7 (11.5)
  Hour 21 | -10.5 (12.3) | -8.6 (14.3) | -8.4 (12.1) | -15.1 (9.4)
  Hour 22 | -10.9 (11.3) | -10 (14.6) | -10.2 (13.5) | -15.2 (10.2)
  Hour 23 | -10 (11.8) | -14 (13.8) | -10 (12.5) | -14.3 (8.5)
  Hour 24 | -9.7 (9.8) | -13.6 (11.2) | -13.2 (13.8) | -14.4 (12.2)

41. Secondary Outcome: Change From Baseline in ABPM 24-hour Mean DBP
Description: Observed results for mod-sev patients - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 41 | 41 | 46 | 41
mmHg | -11 (7.7) | -13.6 (8) | -13.6 (7.1) | -15.3 (7)

42. Secondary Outcome: Change From Baseline in ABPM 24-hour Mean SBP
Description: Observed results for mod-sev patients - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 41 | 41 | 46 | 41
mmHg | -16.7 (11.3) | -20.8 (14.1) | -20.9 (11) | -22.7 (9.9)

43. Secondary Outcome: Orthostatic Change in Trough Cuff Mean DBP
Description: Calculated as seated minus standing for mod-sev patients - key combination therapies
Time Frame: Week 8
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 102 | 87 | 99 | 88
mmHg | 2.5 (5.1) | 2 (5.7) | 1.4 (5.3) | 1.6 (4.5)

44. Secondary Outcome: Orthostatic Change in Trough Cuff Mean SBP
Description: Calculated as seated minus standing for mod-sev patients - key combination therapies
Time Frame: Week 8
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 102 | 87 | 99 | 88
mmHg | 0 (7.1) | 1.4 (8.1) | 0.1 (6.9) | 1.1 (6.3)

45. Secondary Outcome: Change From Baseline in Seated Trough Pulse Rate
Description: Observed results for mod-sev patients - key combination therapies
Time Frame: Up to 8 weeks (LOCF)
Population: The full analysis set relating to the in-clinic trough pulse rate measurements included all treated patients that had at least one in-clinic pulse rate measurement following treatment with target therapy and were identified as having moderate or severe hypertension at baseline (FAS-TC-MS).
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10)
Number analyzed (Participants) | 108 | 96 | 106 | 100
bpm | 0.5 (8.8) | 0 (9) | 2.5 (9.2) | -1.9 (8.9)

46. Secondary Outcome: Clinical Relevant Abnormalities for Laboratory Parameters and Electrocardiogram (ECG)
Description: Clinical relevant abnormalities for laboratory parameters and Electrocardiogram (ECG). New abnormal findings or worsening of baseline conditions were reported as Adverse Events related to treatment (cardiac disorders and investigations).
Time Frame: 8 weeks
Population: Treated set
Measure: Number; unit: percentage of participants
Groups:
- Telmisartan Monotherapy: Telmisartan 20/40/80mg tablet, QD in morning
- Amlodipine Monotherapy: encapsulated Amlodipine 2.5/5 mg capsule or 2 x 5mg capsules, QD in morning
- Combination Therapy: Telmisartan 20/40/80mg tablet plus 2.5/5 mg capsule or 2 x 5mg capsules, QD in morning
Arm/Group | Placebo (Pl) | Telmisartan Monotherapy | Amlodipine Monotherapy | Combination Therapy
Number analyzed (Participants) | 46 | 307 | 319 | 789
percentage of participants
  Alanine aminotransferase increased | 0.0 | 0.3 | 0.0 | 0.1
  Aspartate aminotransferase increased | 0.0 | 0.3 | 0.0 | 0.1
  Blood potassium increased | 0.0 | 0.3 | 0.0 | 0.0
  Electrocardiogram QT shortened | 0.0 | 0.0 | 0.3 | 0.0
  Electrocardiogram T wave abnormal | 0.0 | 0.0 | 0.3 | 0.1
  Electrocardiogram repolarisation abnormality | 0.0 | 0.0 | 0.0 | 0.1
  Heart rate irregular | 0.0 | 0.0 | 0.3 | 0.0
  QRS axis abnormal | 0.0 | 0.0 | 0.3 | 0.0
  Atrioventricular block first degree | 0.0 | 0.0 | 0.0 | 0.3
  Left atrial dilatation | 0.0 | 0.0 | 0.0 | 0.1
  Myocardial ischaemia | 0.0 | 0.1 | 0.0 | 0.0
  Palpitation | 0.0 | 0.0 | 0.6 | 0.1
  Sinus bradycardia | 0.0 | 0.0 | 0.0 | 0.1

ADVERSE EVENTS:
Arm/Group | PLACEBO | Telmisartan 20 mg (T20) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg (T40) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg (T80) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/42 | 0/44 | 0/46 | 0/44 | 0/130 | 0/47 | 0/143 | 0/129 | 1/135 | 2/48 | 2/146 | 0/142 | 1/50 | 1/140 | 0/129
Other Adverse Events (participants affected / at risk) | 6 | 5 | 4 | 5 | 6 | 13 | 3 | 9 | 13 | 5 | 1 | 10 | 23 | 2 | 10 | 29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=46) | Telmisartan 20 mg (T20) (N=42) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) (N=44) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) (N=46) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) (N=44) | Telmisartan 40 mg (T40) (N=130) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) (N=47) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) (N=143) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) (N=129) | Telmisartan 80 mg (T80) (N=135) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) (N=48) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) (N=146) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) (N=142) | Amlodipine 2.5 mg (A2.5) (N=50) | Amlodipine 5 mg (A5) (N=140) | Amlodipine 10 mg (A10) (N=129)
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | PLACEBO | Telmisartan 20 mg (T20) | Telmisartan 20 mg Plus Amlodipine 2.5 mg (T20+A2.5) | Telmisartan 20 mg Plus Amlodipine 5 mg (T20+A5) | Telmisartan 20 mg Plus Amlodipine 10 mg (T20+A10) | Telmisartan 40 mg (T40) | Telmisartan 40 mg Plus Amlodipine 2.5 mg (T40+A2.5) | Telmisartan 40 mg Plus Amlodipine 5 mg (T40+A5) | Telmisartan 40 mg Plus Amlodipine 10 mg (T40+A10) | Telmisartan 80 mg (T80) | Telmisartan 80 mg Plus Amlodipine 2.5 mg (T80+A2.5) | Telmisartan 80 mg Plus Amlodipine 5 mg (T80+A5) | Telmisartan 80 mg Plus Amlodipine 10 mg (T80+A10) | Amlodipine 2.5 mg (A2.5) | Amlodipine 5 mg (A5) | Amlodipine 10 mg (A10)
Chest pain (General disorders) | 1/46 | 3/42 | 0/44 | 0/46 | 0/44 | 2/130 | 0/47 | 1/143 | 1/129 | 0/135 | 0/48 | 1/146 | 0/142 | 0/50 | 0/140 | 1/129
Oedema peripheral (General disorders) | 0/46 | 0/42 | 1/44 | 2/46 | 5/44 | 1/130 | 0/47 | 2/143 | 7/129 | 1/135 | 1/48 | 3/146 | 16/142 | 1/50 | 1/140 | 23/129
Headache (Nervous system disorders) | 5/46 | 3/42 | 3/44 | 4/46 | 2/44 | 11/130 | 3/47 | 7/143 | 5/129 | 4/135 | 0/48 | 6/146 | 7/142 | 2/50 | 9/140 | 7/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.